CLINICAL TRIAL: NCT00072059
Title: An Open Label, Randomized, Multicenter, Phase II Study To Determine Hemoglobin Dose Response, Safety And Pharmacokinetic Profile Of Ro 50-3821 Given Subcutaneously Once Weekly Or Once Every 3 Weeks To Anemic Patients With Stage IIIB or IV Non-Small Cell Lung Carcinoma Receiving Antineoplastic Therapy
Brief Title: Ro 50-3821 in Treating Anemia in Patients Receiving Antineoplastic Therapy for Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: ROCHE-NA17101; UCLA-0303085; CDR0000335429 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2005-01

CONDITIONS: Anemia; Lung Cancer
Keywords: anemia; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Anemia; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — continuous erythropoietin receptor activator

INTERVENTIONS:
Biological: methoxy polyethylene glycol epoetin beta

SUMMARY:
RATIONALE: Ro 50-3821 may stimulate red blood cell production and treat anemia in patients who are receiving antineoplastic therapy for non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying six different regimens of Ro 50-3821 to compare how well they work in treating anemia in patients who are receiving antineoplastic therapy for stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the hemoglobin dose response of anemic patients with stage IIIB or IV non-small cell lung cancer receiving antineoplastic therapy treated with 6 different regimens of Ro 50-3821.

Secondary

* Compare the safety profile of these regimens in these patients.
* Compare the pharmacokinetic profile of these regimens in these patients.
* Determine additional pharmacodynamic characteristics of these regimens in these patients.

OUTLINE: This is a randomized, open-label, parallel, multicenter study. Patients are randomized to 1 of 6 treatment arms. In all arms, patients begin study therapy on the first day of a course of antineoplastic therapy.

* Arm I: Patients receive a lower dose of Ro 50-3821 subcutaneously (SC) once weekly.
* Arm II: Patients receive a medium dose of Ro 50-3821 SC once weekly.
* Arm III: Patients receive a higher dose of Ro 50-3821 SC once weekly.
* Arm IV: Patients receive a lower dose of Ro 50-3821 SC once every 3 weeks.
* Arm V: Patients receive a medium dose of Ro 50-3821 SC once every 3 weeks.
* Arm VI: Patients receive a higher dose of Ro 50-3821 SC once every 3 weeks. In all arms, treatment continues for 12 weeks in the absence of unacceptable toxicity.

Patients are followed at 1 week.

PROJECTED ACCRUAL: A total of 210 patients (35 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIB or IV
* Currently receiving first- or second-line antineoplastic therapy (must be scheduled to receive therapy during the 12 weeks of study therapy)

  * Antineoplastic therapy may include single agent or combination chemotherapy, corticosteroids, or a combination of these agents
* Hemoglobin no greater than 11 g/dL

  * Transfusion independent
* No known primary or metastatic CNS malignancy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* See Disease Characteristics
* Platelet count 50,000-500,000/mm^3
* No functional iron deficiency* (e.g., transferrin saturation less than 20% OR serum ferritin less than 100 ng/mL)
* No known hemolysis NOTE: *Concurrent iron supplementation to correct deficiency allowed

Hepatic

* Not specified

Renal

* Creatinine no greater than 2.5 mg/dL

Cardiovascular

* No clinically significant hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix
* No acute or chronic bleeding requiring therapy within the past 3 months (e.g., patients with anemia caused by gastrointestinal bleeding)
* No known cyanocobalamin deficiency
* No known folic acid deficiency
* No acute infection or inflammatory disease (C-reactive protein greater than 50 mg/L)
* No known resistance to epoetin administration
* No newly diagnosed (i.e., within the past 6 months) or uncontrolled epilepsy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 8 weeks since prior recombinant human erythropoietin therapy or any other erythropoiesis-stimulating drugs

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 4 weeks since prior red blood cell transfusion
* More than 30 days since prior investigational drugs or regimens
* No prior enrollment and randomization to this study
* No other concurrent investigational drugs or regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States